CLINICAL TRIAL: NCT04340791
Title: Effectiveness of Information-based Versus Structural Interventions on Food Choices by Socioeconomic Position: a Randomized Controlled Trial in an Experimental Online Supermarket
Brief Title: Increased Proportion of Lower Energy Density Items vs. Nutritional Labelling at an Online Supermarket
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Eric Robinson, Principal Investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 803194 1B3
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Diet, Healthy; Food Selection
Keywords: availability; labelling; food choice; socio-economic position
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Default proportion & no labelling (No Intervention): No intervention:
  Default proportion condition (33% lower energy density items - 67% higher energy density items). Lower energy density items will be defined as lower ED ≤ median of ED distribution within a food category.
  No labelling.
- Default proportion & labelling (Experimental): When energy density of a food item ≤ median of energy density distribution within a food category, "healthier choice" badges will be added to the food item pictures on the online supermarket. Instructions will introduce the badges to the participants as "In the online supermarket, the green tick allows you to see which products (e.g. muesli) in each product category (e.g. cereals) are healthier choices with fewer calories per gram than most other products in the same category."
  Interventions: Behavioral: Labelling
- Increased proportion & no labelling (Experimental): The proportion of lower energy density items vs. higher energy density items will be reversed (67% lower - 33% higher) relative to the default proportion condition (33% lower - 67% higher). Lower energy density items will be defined as lower ED ≤ median of ED distribution within a food category.
  Interventions: Behavioral: Increased proportion of lower energy density items
- Increased proportion & labelling (Experimental): The proportion of lower energy density items vs. higher energy density items will be reversed (67% lower - 33% higher) relative to the default proportion condition (33% lower - 67% higher). Lower energy density items will be defined as lower ED ≤ median of ED distribution within a food category.
  When energy density of a food item ≤ median of energy density distribution within a food category, "healthier choice" badges will be added to the food item pictures on the online supermarket. Instructions will introduce the badges to the participants as "In the online supermarket, the green tick allows you to see which products (e.g. muesli) in each product category (e.g. cereals) are healthier choices with fewer calories per gram than most other products in the same category."
  Interventions: Behavioral: Increased proportion of lower energy density items; Behavioral: Labelling

INTERVENTIONS:
Behavioral: Increased proportion of lower energy density items — The proportion of lower energy density vs. higher energy density items will be reversed (67% lower - 33% higher) relative to the default proportion condition (D and DL) (33% lower - 67% higher). Lower energy density items will be defined as lower energy density ≤ median of energy density distribution within a food category.
  Arms: Increased proportion & labelling; Increased proportion & no labelling
Behavioral: Labelling — When energy density of an item ≤ median of ED distribution within a food category, "healthier choice" badges will be added to the food item pictures on the online supermarket. Instructions when logging-into the platform will introduce the badges to the participants: "In the online supermarket, the green tick allows you to see which products (e.g. muesli) in each product category (e.g. cereals) are healthier choices with fewer calories per gram than most other products in the same category."
  Arms: Default proportion & labelling; Increased proportion & labelling

SUMMARY:
This study will be a 2x2 randomised controlled trial with information-based intervention (no labelling / labelling) and structural intervention (default proportion / increased proportion of lower energy density food items) as between-subject factors and energy density (kcal/g) of food purchases during an online supermarket-shopping task as dependent variable. This study will use an online supermarket platform developed to mimic an online supermarket website and participants will be asked to complete a shopping task using a pre-determined shopping list of 10 items.

DETAILED DESCRIPTION:
See attached protocol documents.

ELIGIBILITY:
Inclusion Criteria:

* United Kingdom residents
* Aged ≥ 18 years
* Fluent in English
* Have access to a computer and Internet
* Responsible for a substantial proportion of household grocery shopping

Exclusion Criteria:

* Unable to provide informed consent and to comply with the study requirements
* Any dietary restriction (vegetarian, vegan, gluten-free, sugar-free, dairy or lactose free, food allergy, other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-05-13 (Actual)

PRIMARY OUTCOMES:
Mean ED of the food items purchased (kcal/100g) | 20 minutes (the time frame denotes time taken to make the food shopping task online and there is no follow up)
  Calculated as the sum of the energy of the purchased items (kcal) divided by the sum of their weight (g) and multiplied by 100.

SECONDARY OUTCOMES:
Total energy of the food items purchased (kcal) | 20 minutes (the time frame denotes time taken to make the food shopping task online and there is no follow up)
  Calculated as the sum of the energy of the purchased items (kcal)
Energy from total sugar (% of total energy) | 20 minutes (the time frame denotes time taken to make the food shopping task online and there is no follow up)
  Calculated as the percentage of total energy of the purchased items from total sugar
Energy from saturated fatty acids (SFA) (% of total energy) | 20 minutes (the time frame denotes time taken to make the food shopping task online and there is no follow up)
  Calculated as the percentage of total energy of the purchased items from SFA
Salt content (g/100g) | 20 minutes (the time frame denotes time taken to make the food shopping task online and there is no follow up)
  Calculated as the sum of the salt content of the purchased items (g) divided by the sum of their weight (g) and multiplied by 100.
Proportion of lower energy density food items in the basket of foods purchased | 20 minutes (the time frame denotes time taken to make the food shopping task online and there is no follow up)
  Lower energy density items will be defined as ≤ median of energy density distribution within a food category
Cost (GPB) | 20 minutes (the time frame denotes time taken to make the food shopping task online and there is no follow up)
  Calculated as the sum of the prices of the purchased items

OTHER OUTCOMES:
Validity | 5 minutes (the time frame denotes time taken to fill in the debriefing questionnaire and there is no follow up)
  Mean of item "I would normally buy [the 10 items on the shopping list]" for all the food items coded as: 1 = Never; 2 = Very rarely; 3 = Rarely; 4 = Occasionally; 5 = Frequently; 6 = Very frequently.
Kcal influence | 5 minutes (the time frame denotes time taken to fill in the debriefing questionnaire and there is no follow up)
  Answer to the item "The choices I made during online shopping were influenced by how many calories I thought were in the options available." coded as: 1 = Strongly disagree; 2 = Disagree; 3 = Slightly disagree; 4 = Neutral; 5 = Slightly agree; 6 = Agree; 7 = Strongly agree

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Shared on the Open Science Framework
Supporting Information: Study Protocol, SAP, ICF
Time Frame: On publication, indefinitely
Access Criteria: Open website
URL: https://osf.io/kq9c8/

REFERENCES:
- Available data/document: Study Protocol — https://osf.io/kq9c8/
- Available data/document: Statistical Analysis Plan — https://osf.io/kq9c8/
- Available data/document: Informed Consent Form — https://osf.io/kq9c8/
- Available data/document: Individual Participant Data Set — https://osf.io/kq9c8/ — When results will be published

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT04340791/Prot_SAP_ICF_000.pdf